CLINICAL TRIAL: NCT06976528
Title: Understanding the Associations Between Romantic Relationship Conflict, Psychophysiological Responding and Alcohol Misuse Among Emerging Adults
Status: Recruiting | Type: Observational
Sponsor: New York University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20237802; 5K23AA030328 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Heavy Episodic Drinking
Keywords: couples; emerging adults; young adults; binge drinking; alcohol use; conflict
MeSH Terms: conditions — Binge Drinking; Alcohol Drinking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emerging Adults (EA) engage in heavy episodic drinking (HED) at a greater quantity and frequency than any other time in their lives, which may lead to significant short- and long-term consequences. Although much is known about the influence of peers in EA alcohol use, there is a dearth of research examining the ways in which romantic partners influence EA drinking behaviors. The proposed study bridges a crucial gap in the existing literature by examining behavioral and physiological risk and resilience factors in the acute link between EA relationship conflict and alcohol consumption. EA couples will engage in two conflict resolution tasks interspersed with two puzzle tasks and two alcohol administration procedures. Because high frequency heart rate variability (HF-HRV) is associated with alcohol use and emotion regulation during stressful experiences, HF-HRV and other physiological data will be collected throughout the laboratory procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-29 years old
2. Must be in a committed romantic relationship of at least 3 months duration
3. Must report at least 2 HED episodes in the past 30 days (5 or more drinks within 2 hours for males, 4 or more drinks within 2 hours for females)
4. Must self-report that they have - on at least three occasions during the past year - consumed a quantity of alcohol that is equal to or greater than the standard dose administered for their weight in the laboratory

Exclusion Criteria:

1. Meeting DSM-5 criteria for a history of or current neurological, psychotic, or bipolar disorders
2. History of self-reported head trauma requiring medical treatment
3. Body weight exceeding 250 pounds
4. Current enrollment in treatment or seeking treatment for a substance or alcohol use disorder
5. Current suicidal or homicidal intent
6. Serious cardiovascular health conditions (e.g. pacemaker, cardiac arrhythmia, hypertension) that may alter normative cardiac functioning
7. Treatment on medications such as lithium, methadone, alpha or beta blockers or cholinergic/anticholinergic medications likely to confound normative cardiovascular responding or response to alcohol administration. Stimulant or benzodiazepine medication use is permissible provided participants do not take medication on the day of study participation
8. Severe and/or unilateral physical IPV with your current partner at any time
9. Sexual IPV with current partner at any time
10. Fear of current partner
11. Pregnancy or breastfeeding
12. Severe Alcohol Use Disorder (as defined by the DSM-5)
13. Current diagnosis of anorexia or bulimia

Ages: 21 Years to 29 Years | Sex: All
Age Groups: Adult
Study Population: Emerging adults in couples in the NYC area
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | ~20 minutes
  Amount of alcohol consumed during the study

SECONDARY OUTCOMES:
High frequency heart rate variability (HF-HRV) | ~3 hours
  High frequency heart rate variability (HF-HRV) is a neurally-derived measure of parasympathetic activity that may partially explain the association between stressful relationship conflict and alcohol misuse. HF-HRV is a measure of the variability in interbeat intervals, or the time in between beats of the heart.

CONTACTS AND LOCATIONS:
Locations (1):
- 386 Park Avenue South, New York, New York, United States